CLINICAL TRIAL: NCT06556979
Title: Carotid Artery Stenosis and Ischemic Cerebrovascular Events After Radiotherapy in Patients With Head and Neck Cancer
Acronym: RT-CASinHNC
Status: Completed | Type: Observational
Sponsor: Chulabhorn Royal Academy (Other)
Responsible Party: Principal Investigator, Nawaphan Taengsakul, Principal Investigator, Chulabhorn Royal Academy
Other Study IDs: EC 048/2565
Record Dates: First submitted 2024-08-08; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Carotid Artery Stenosis; Head and Neck Cancer; Radiation Therapy; Transient Ischemic Attack; Ischemic Stroke
Keywords: Carotid artery stenosis; Head and neck cancer; Radiation therapy; Transient ischemic attack; Ischemic stroke; Thailand
MeSH Terms: conditions — Carotid Stenosis; Head and Neck Neoplasms; Ischemic Attack, Transient; Ischemic Stroke | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HNC patient who recieve RT: Reviewing medical record of all patiented who receive radiotherapy and focusing in ischemic cerebrovascular event and carotid artery stenosis. We categorized the patiented to 3 group : no carotid artery stenosis, seen carotid artery stenosis and seen significant carotid artery stenosis and find the risk factor of preexisting carotid artery stenosis before RT
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — Review imaging and medical record of head and neck cancer patient who recieve radiotherpy to find out the incidence of ischemic cerebrovascular event and carotid artery stenosis. The risk factor that influence new carotid artery stenosis was claculated

SUMMARY:
The study had a cross-sectional design and included patients with HNC involving the oral cavity, pharynx, larynx, nasal cavity, or salivary glands who recieve RT.

the investigators obtained information on their clinical and tumor characteristics and their treatment from the clinical records. Data on risk factors for atherosclerosis, medications used, and radiotherapy were also collected.

Images were analyzed to determine the timing of development of CAS, identify significant (>50%) CAS using the North American Symptomatic Carotid Endarterectomy Trial criteria, and calculate the total plaque score (TPS) and wall thickness.

The purpose of this study was to determine the incidence of ICVE and of CAS in patients who receive radiotherapy for HNC and the risk factors for CAS.

DETAILED DESCRIPTION:
The study had a cross-sectional design and included 907 patients with HNC involving the oral cavity, pharynx, larynx, nasal cavity, or salivary glands. The study was approved by the Chulabhorn Institutional Ethics Committee for Human Research (approval number 048/2565). All patients underwent radiotherapy to the head and neck region between February 2011 and June 2022 with or without surgical resection and were investigated by computed tomography (CT) before and after radiotherapy. Patients with lymphoma and those with previous treatment for CAS or radiotherapy for other diseases were excluded. We obtained information on patient background factors, tumor characteristics, and treatment from the medical records. Risk factors for atherosclerosis, including hypertension, dyslipidemia, diabetes mellitus, coronary artery disease, peripheral arterial disease, and cigarette smoking, were identified. Baseline laboratory data, including hemoglobin A1C, fasting blood sugar, lipid profile, serum creatinine level, and estimated glomerular filtration rate, were obtained, as was information on treatment, including antiplatelet agents, statins, angiotensin-converting enzyme inhibitors (ACEIs), calcium channel blockers (CCBs), and anticoagulants. The type and stage of HNC, indication for radiotherapy, type of radiotherapy, total cumulative dose, and number of courses were also recorded. Unfortunately, the laboratory data were incomplete in many cases, so could not be subjected to statistical analysis. Follow-up was continued until loss to follow-up, death, or the end of 2023, whichever came first. Moreover, full written informed consent was obtained from the patient for publication of this article. Confidentiality of the data was secured by assigning of a code for each patient record. Images were analyzed to determine the timing of development of CAS, identify significant (>50%) CAS using the North American Symptomatic Carotid Endarterectomy Trial criteria, and calculate the total plaque score (TPS) and wall thickness. The carotid vessels were divided into the common carotid artery (CCA), carotid bulb, internal carotid artery (ICA), and external carotid artery (ECA). The bulb was defined as the portion of the artery 1 cm caudally to 1 cm cranially from the point where the CCA divided into the ICA and ECA. The right and left carotid artery systems were each divided into the following five segments: proximal CCA (≥20 mm proximal to bulb), distal CCA (<20 mm proximal to bulb), carotid bulb, ICA. and ECA. Each segment was graded as follows: 0, normal or no detectable plaque; 1, plaque occupying <30% of vessel diameter; 2, plaque occupying 30%-49% of vessel diameter; 3, plaque occupying 50%-69% of vessel diameter; 4, plaque occupying 70%-99% of vessel diameter; and 5, 100% occlusion of vessel diameter by plaque. The carotid plaque score was obtained for each patient by summing the scores obtained for the five arterial segments in both carotid arteries. Wall thickness and degree of CAS were measured in the five segments of the carotid artery at baseline and during follow-up. Differences in these values were calculated. CT was performed at least twice. The initial CT scan was performed within 2 months before initiation of radiotherapy and follow-up CT was performed 1 month after completing radiotherapy. In cases with multiple follow-up CT scans, the last scan was used to evaluate post-radiation change. The 1-year follow-up CT scan was also examined. All baseline and follow-up measurements were made by a vascular surgeon who was blinded to the clinical data.

ELIGIBILITY:
Inclusion Criteria:

* All patients underwent radiotherapy to the head and neck region between February 2011 and June 2022 with or without surgical resection and were investigated by computed tomography (CT) before and after radiotherapy.

Exclusion Criteria:

* Patients with lymphoma and those with previous treatment for CAS or radiotherapy for other diseases were excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with HNC involving the oral cavity, pharynx, larynx, nasal cavity, or salivary glands.
Sampling Method: Non-Probability Sample
Enrollment: 907 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Incidence of ischemic cerebrovascular event after radiotherapy. (Percentage of partcipants who developed ischemic stroke or transient ischemic attack following completion of radiotherapy in all participants) | 5 years
  The cumulative incidence of ischemic cerbrovascular event including ischemic stroke or transient ischemic attack in the anterior circulation in HNC patient who receive radiotherapy in 5 years

SECONDARY OUTCOMES:
The risk factors that were identified to influence development of new carotid artery stenosis | through study completion, an average of 1 year
  The risk factors that were identified to influence development of new carotid artery stenosis from the first imaging to last imaging. The investigator assessed the number of patient who develop new carotid artery stenosis after radiotherapy. Carotid artery stenosis was measure by NASCET criteria : % ICA stenosis = (1 - [narrowest ICA diameter/diameter normal distal cervical ICA]) x 100
Incidence of carotid artery stenosis at 12, 24, and 36 months after radiotherapy (Percentage of partcipants who develop carotid artery stenosis) | 12, 24, 36 months
  The cumulative incidence of carotid artery stenosis was calculated after radiotherapy. The investigator assessed the number of patient who develop new carotid artery stenosis after radiotherapy. Carotid artery stenosis was measure by NASCET criteria : % ICA stenosis = (1 - [narrowest ICA diameter/diameter normal distal cervical ICA]) x 100

CONTACTS AND LOCATIONS:
Overall Officials: Nawaphan Taengsakul Taengsakul, MD, Principal Investigator — Chulabhorn Royal Academy
Locations (1):
- Department of Surgery, Chulabhorn Hospital, Princess Srisavangavadhana College of Medicine, Chulabhorn Royal Academy, Bangkok, Thailand, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided